CLINICAL TRIAL: NCT04758728
Title: The Role of Adrenaline in the Reduction of Subcutaneous Ecchymoses and Hematomas and in the Improvement of the Quality of Life of Patients After Classic Great Saphenous Vein Stripping
Brief Title: Adrenaline Reduces Ecchymoses and Hematomas and Improves Quality of Life After Classic Saphenous Vein Stripping
Acronym: ARESQOLSAVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junior Doctors Network-Hellas (Other)
Collaborators: General Hospital of Rhodes Andreas Papandreou (Other Government); Hellenic Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Roditis, MD, MSc, Chief Resident, JDN-Hellas Board Chairperson, Junior Doctors Network-Hellas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARES-QOL-SAVES
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Venous Insufficiency (Chronic)(Peripheral); Venous Reflux; Venous Insufficiency of Leg; Venous Stasis; Venous Disease; Subcutaneous Haematoma; Ecchymosis; Bruising
Keywords: great saphenous vein; saphenectomy; saphenous vein stripping; ecchymosis; haematoma; adrenaline; epinephrin; hemostasis; chronic venous insufficiency; venous reflux; venous disease
MeSH Terms: conditions — Venous Insufficiency; Varicose Ulcer; Ecchymosis; Contusions; Hematoma | interventions — Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Group A - great saphenous vein stripping with local adrenaline use for hemostasis
  Interventions: Procedure: Great saphenous vein stripping and varicectomies; Drug: Epinephrine Topical
- Group B (Sham Comparator): Group B - great saphenous vein stripping with local normal saline use for hemostasis
  Interventions: Procedure: Great saphenous vein stripping and varicectomies; Drug: normal saline
- Group C (Sham Comparator): Group C - great saphenous vein stripping with traditional hemostatic practice
  Interventions: Procedure: Great saphenous vein stripping and varicectomies

INTERVENTIONS:
Procedure: Great saphenous vein stripping and varicectomies — Removal of the great saphenous vein (partially - from just below the knee up to the saphenofemoral junction) by two 3cm skin and subcutaneous fat incisions and the introduction of a conventional vein stripper device, under general or epidural/regional anesthesia. Removal of varicose veins of the lower limb by 0,5cm skin incisions and the use of a conventional phlebectomy stainless steel hook. Mechanical hemostasis by direct compression of the thigh for 10 minutes.
  Other Names: Saphenectomy
Drug: Epinephrine Topical — Use of epinephrine/adrenaline solution 1:1000 topically
  Other Names: Adrenaline solution 1:1000 topical/local use
  Arms: Group A
Drug: normal saline — Use of normal saline solution NaCl 0,9% topically
  Other Names: NaCl 0,9% topical/local use
  Arms: Group B

SUMMARY:
Aim of the present study is to investigate the efficiency of adrenaline (epinephrine) used locally in reducing and avoiding post-operative formation of subcutaneous ecchymoses and hematomas, in comparison with traditional practice of hemostasis, and to assess improvement in the quality of life of subjects undergoing classic great saphenous vein stripping, who received or did not receive adrenaline as a local hemostatic.

DETAILED DESCRIPTION:
Introduction Quality of life of subjects undergoing classic great saphenous vein stripping is analogous of the gravity of subcutaneous ecchymoses and hematomas formation, as a result of surgical interventions during open surgery, when the great saphenous vein is being removed. Adrenaline (epinephrine) is a potent vasoconstrictor, whose local hemostatic ability has already been documented and applied in many medical specialties. Aim of the present study to investigate the efficiency of adrenaline (epinephrine) used locally in reducing and avoiding post-operative formation of subcutaneous ecchymoses and hematomas, in comparison with traditional practice of hemostasis, and to assess improvement in the quality of life of subjects undergoing classic great saphenous vein stripping, who received or did not receive adrenaline as a local hemostatic.

Material-Methods 40 subjects diagnosed with chronic venous insufficiency (CVI) and/or varicose veins of the lower limbs of varied clinical gravity (CEAP classification II & III), admitted in the department of Vascular Surgery for open surgical management, i.e. great saphenous vein stripping +/- removal of varicosities, will be enrolled after signing an informed consent for their participation in the study. They will be then randomized into 3 separate groups: Group A - great saphenous vein stripping with local adrenaline use for hemostasis Group B - great saphenous vein stripping with local normal saline use for hemostasis Group C - great saphenous vein stripping with traditional hemostatic practice Study subjects will be followed-up after surgery, and in each group measurement of ecchymoses (small 2-5mm2 and large >5mm2) and hematomas (medium 0,2-1cm and large >1cm) will be performed by using ImageJ software after digital high-resolution photographing on 1st, 8th and 14th post-operative days. Quality of life of subjects will be assessed pre-operatively and 1 month post-operatively, by using SF-36 and CIVIQ-2 questionnaires for QoL in CVI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* CVI CEAP Class II or III
* Informed consent signed

Exclusion Criteria:

* Age <18 or >80 years
* CVI CEAP Class I or IV (venous ulcers)
* Allergy to adrenaline history
* No informed consent signed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2016-05-14 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
Subcutaneous ecchymoses number 1d-postop | 24 hours post-operatively
  The absolute number of subcutaneous ecchymoses on the operated limb on 1st post-operative day
Subcutaneous ecchymoses number 8d-post-op | 192 hours post-operatively
  The absolute number of subcutaneous ecchymoses on the operated limb on 8th post-operative day
Subcutaneous ecchymoses number 14d-post-op | 336 hours post-operatively
  The absolute number of subcutaneous ecchymoses on the operated limb on 14th post-operative day
Subcutaneous hematomas number 1d-postop | 24 hours post-operatively
  The absolute number of subcutaneous hematomas in the operated limb on 1st post-operative day
Subcutaneous hematomas number 8d-postop | 192 hours post-operatively
  The absolute number of subcutaneous hematomas in the operated limb on 8th post-operative day
Subcutaneous hematomas number 14d-postop | 336 hours post-operatively
  The absolute number of subcutaneous hematomas in the operated limb on 14th post-operative day
Subcutaneous ecchymoses total area 1d-postop | 24 hours post-operatively
  The total area in mm2 of subcutaneous ecchymoses in the operated limb on 1st post-operative day
Subcutaneous ecchymoses total area 8d-postop | 192 hours post-operatively
  The total area in mm2 of subcutaneous ecchymoses in the operated limb on 8th post-operative day
Subcutaneous ecchymoses total area 14d-postop | 336 hours post-operatively
  The total area in mm2 of subcutaneous ecchymoses in the operated limb on 14th post-operative day
Subcutaneous hematomas total area 1d-postop | 24 hours post-operatively
  The total area in mm2 of subcutaneous hematomas in the operated limb on 1st post-operative day
Subcutaneous hematomas total area 8d-postop | 192 hours post-operatively
  The total area in mm2 of subcutaneous hematomas in the operated limb on 8th post-operative day
Subcutaneous hematomas total area 14d-postop | 336 hours post-operatively
  The total area in mm2 of subcutaneous hematomas in the operated limb on 14th post-operative day
QoL-SF36 preop | 24 hours pre-operatively
  Quality of life assessment based on the 36-Item Short Form Survey (SF-36) questionnaire preoperatively. It is an often-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study. It taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The eight scaled scores, which are the weighted sums of the questions in their section are directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
QoL-SF36 1month-postop | 30 days post-operatively
  Quality of life assessment based on the 36-Item Short Form Survey (SF-36) questionnaire 30 days post-operatively. It is an often-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study. It taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The eight scaled scores, which are the weighted sums of the questions in their section are directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
QoL-CIVIQ2 preop | 24 hours pre-operatively
  Quality of life assessment based on the ChronIc Venous Insufficiency quality of life Questionnaire version 2 (CIVIQ-2) questionnaire preoperatively. The CIVIQ was developed and validated (relevance, acceptability, reliability, construct validity, and sensitivity) by French researchers in 1996. The CIVIQ is a 20-item self-reported instrument that includes four categories of questions: physical (4 items), psychological (9 items), social (4 items), and pain (3 items). Its score ranges from 0, the worst score, to 100, the best. There are five possible answers (from 1 to 5) to describe each symptom and the sensation of discomfort. The second version, the CIVIQ-2 (where 2 denotes the second draft of the same questionnaire), provides a global score covering all aspects of the questionnaire and weighs the categories equally.
QoL-CIVIQ2 1month post-op | 30 days post-operatively
  Quality of life assessment based on the CIVIQ-2 questionnaire 1 month post-operatively. Quality of life assessment based on the ChronIc Venous Insufficiency quality of life Questionnaire version 2 (CIVIQ-2) questionnaire preoperatively. The CIVIQ was developed and validated (relevance, acceptability, reliability, construct validity, and sensitivity) by French researchers in 1996. The CIVIQ is a 20-item self-reported instrument that includes four categories of questions: physical (4 items), psychological (9 items), social (4 items), and pain (3 items). Its score ranges from 0, the worst score, to 100, the best. There are five possible answers (from 1 to 5) to describe each symptom and the sensation of discomfort. The second version, the CIVIQ-2 (where 2 denotes the second draft of the same questionnaire), provides a global score covering all aspects of the questionnaire and weighs the categories equally.

SECONDARY OUTCOMES:
HCT preop | 24 hours pre-operatively
  Hematocrit (HCT) measured pre-operatively, in percentage (%).
HCT postop | 24 hours post-operatively
  Hematocrit (HCT) measured post-operatively, in percentage (%).
Hgb preop | 24 hours pre-operatively
  Hemoglobin (Hgb) measured pre-operatively, in mg/dL.
Hgb postop | 24 hours post-operatively
  Hemoglobin (Hgb) measured post-operatively, in mg/dL.
WBC preop | 24 hours pre-operatively
  White blood cells (WBC) count measured pre-operatively, in K/mcL.
WBC postop | 24 hours post-operatively
  White blood cells (WBC) count measured post-operatively, in K/mcL.
PLT preop | 24 hours pre-operatively
  Platelet count (PLT) measured pre-operatively, in K/mcL.
PLT postop | 24 hours post-operatively
  Platelet count (PLT) measured post-operatively, in K/mcL.
FIB preop | 24 hours pre-operatively
  Fibrinogen (FIB) measured pre-operatively, in mg/dL.
FIB postop | 24 hours post-operatively
  Fibrinogen (FIB) measured post-operatively, in mg/dL.
ESR preop | 24 hours pre-operatively
  Erythrocyte sedimentation rate on the 1st hour, measured pre-operatively, in millimeters (mm).
ESR postop | 24 hours post-operatively
  Erythrocyte sedimentation rate on the 1st hour, measured post-operatively, in millimeters (mm).
CRP preop | 24 hours pre-operatively
  Serum C-reactive protein (CRP) measured pre-operatively, in mg/L.
CRP postop | 24 hours post-operatively
  Serum C-reactive protein (CRP) measured post-operatively, in mg/L.
Experienced pain preop | 24 hours pre-operatively
  Pain experienced pre-operatively assessed by a numeric rating pain scale (0-10). Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. 0 indicates no pain, 5 moderate and 10 worst possible pain.
Experienced pain 1d-postop | 24 hours post-operatively
  Pain experienced pre-operatively assessed by a numeric rating pain scale (0-10). Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. 0 indicates no pain, 5 moderate and 10 worst possible pain.
Experienced pain 8d-postop | 192 hours post-operatively
  Pain experienced pre-operatively assessed by a numeric rating pain scale (0-10). Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. 0 indicates no pain, 5 moderate and 10 worst possible pain.
Experienced pain 14d-postop | 336 hours post-operatively
  Pain experienced pre-operatively assessed by a numeric rating pain scale (0-10). Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. 0 indicates no pain, 5 moderate and 10 worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Roditis, MD, MSc, Principal Investigator — JDN-Hellas / Department of Vascular Surgery, Hellenic Red Cross Hospital; Dimitrios Mavros, MD, MSc, PhD, Study Chair — Department of Vascular Surgery, Andreas Papandreou General Hospital
Locations (1):
- Department of Vascular Surgery, Andreas Papandreou General Hospital, Rhodes, South Aegean, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuya T, Tada Y, Sato O. A new technique for reducing subcutaneous hemorrhage after stripping of the great saphenous vein. J Vasc Surg. 1992 Sep;16(3):493-4. doi: 10.1016/0741-5214(92)90389-p. No abstract available. PMID 1522653
- [Background] Nisar A, Shabbir J, Tubassam MA, Shah AR, Khawaja N, Kavanagh EG, Grace PA, Burke PE. Local anaesthetic flush reduces postoperative pain and haematoma formation after great saphenous vein stripping--a randomised controlled trial. Eur J Vasc Endovasc Surg. 2006 Mar;31(3):325-31. doi: 10.1016/j.ejvs.2005.08.006. Epub 2005 Oct 19. PMID 16236532
- [Background] Pappa E, Kontodimopoulos N, Niakas D. Validating and norming of the Greek SF-36 Health Survey. Qual Life Res. 2005 Jun;14(5):1433-8. doi: 10.1007/s11136-004-6014-y. PMID 16047519
- [Background] Andreozzi GM, Cordova RM, Scomparin A, Martini R, D'Eri A, Andreozzi F; Quality of Life Working Group on Vascular Medicine of SIAPAV. Quality of life in chronic venous insufficiency. An Italian pilot study of the Triveneto Region. Int Angiol. 2005 Sep;24(3):272-7. PMID 16158038
- [Background] Kim H, Hwang K, Yun SM, Kim DJ. Usage of Epinephrine Mixed With Lidocaine in Plastic Surgery. J Craniofac Surg. 2020 May/Jun;31(3):791-793. doi: 10.1097/SCS.0000000000006156. PMID 32028367